CLINICAL TRIAL: NCT00000437
Title: Nalmefene in Nicotine and Alcohol Dependence
Brief Title: Tobacco Dependence in Alcoholism Treatment (Nicotine Patch/Naltrexone)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Scripps Research Institute (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Barbara J. Mason, Principal Investigator, The Scripps Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIAAAMAS11210; R01AA011210 (NIH)
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Alcoholism; Smoking
MeSH Terms: conditions — Alcoholism; Smoking | interventions — Naltrexone; Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind tablet and patch active study medications, and matched tablet and patch placebos
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Naltrexone Tablet and Nicotine Patch (Experimental)
  Interventions: Drug: Naltrexone Tablet and Nicotine Patch
- Naltrexone Tablet and Placebo Patch (Active Comparator)
  Interventions: Drug: Naltrexone Tablet and Placebo Patch
- Placebo Tablet and Nicotine Patch (Active Comparator)
  Interventions: Drug: Placebo Tablet and Nicotine Patch
- Placebo Tablet and Placebo Patch (Placebo Comparator)
  Interventions: Drug: Placebo Tablet and Placebo Patch

INTERVENTIONS:
Drug: Naltrexone Tablet and Nicotine Patch
  Other Names: Revia and Nicotrol
  Arms: Naltrexone Tablet and Nicotine Patch
Drug: Naltrexone Tablet and Placebo Patch
  Other Names: Revia
  Arms: Naltrexone Tablet and Placebo Patch
Drug: Placebo Tablet and Nicotine Patch
  Other Names: Nicotrol
  Arms: Placebo Tablet and Nicotine Patch
Drug: Placebo Tablet and Placebo Patch
  Arms: Placebo Tablet and Placebo Patch

SUMMARY:
The purpose of this study is to determine the effectiveness of naltrexone (Revia) or matched placebo combined with nicotine patch (Nicotrol) or placebo patch using a 2x2 design in reducing drinking and smoking in patients with both nicotine and alcohol dependence.

DETAILED DESCRIPTION:
Eligible individuals will be randomly assigned to a 12-week trial of a fixed daily dose of either naltrexone (Revia) and nicotine replacement patch or placebos. All individuals will receive weekly coping skills and smoking-cessation behavioral therapy. Followup interviews will be conducted 3 and 6 months after treatment to determine smoking and drinking status and persistence of any dependence symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for alcohol dependence and nicotine dependence.
* Expresses a desire to cut down or stop drinking and smoking.

Exclusion Criteria:

* Currently meets criteria for dependence on substances other than alcohol and nicotine.
* Any history of opiate dependence or evidence of current opiate use.
* Significant medical disorders that will increase potential risk or interfere with study participation.
* Liver function tests more than 3 times normal or elevated bilirubin.
* Females who are pregnant, nursing, or not using a reliable method of birth control.
* Meets criteria for a major psychiatric disorder and is in need of or currently undergoing drug therapy.
* Inability to understand and/or comply with the provisions of the protocol and consent form.
* Treatment with an investigational drug during the previous month.
* Chronic treatment with any narcotic-containing medications during the previous month.
* Sensitivity to drug as evidenced by adverse drug experiences especially with narcotic- containing analgesics or opioid antagonists.
* Current treatment with disulfiram (Antabuse) or nicotine replacement therapy.
* More than 6 weeks of abstinence.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 1997-09-26 (Actual); Primary Completion 2005-09-15 (Actual); Study Completion 2005-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Mason, PhD, Principal Investigator — University of Miam
Locations (1):
- Department of Psychiatry, University of Miami School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No